CLINICAL TRIAL: NCT05449067
Title: Comparison of Efficacy Between Nighttime vs Daytime Peritoneal Dialysis in Non-diabetic Patients: a Randomized, Open-label, Cross-over, Multi-center Clinical Trial
Brief Title: Comparison of Efficacy Between Nighttime and Daytime Peritoneal Dialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Fujian Provincial Hospital (Other); The Affiliated Ganzhou Hospital of Nanchang University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); First People's Hospital of Yulin (Other); Dongguan Tungwah Hospital (Other); Guizhou Provincial People's Hospital (Other); The First People's Hospital of Nanning (Unknown); Tianjin Medical University Second Hospital (Other); Guangzhou First People's Hospital (Other); Fuzhou First General Hospital Affiliated with Fujian Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2022-188
Record Dates: First submitted 2022-06-22; First posted 2022-07-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: End-Stage Kidney Disease; Peritoneal Dialysis
Keywords: Nocturnal Continuous Cyclical Peritoneal Dialysis; Continuous Ambulatory Peritoneal Dialysi; Dialysis Adequacy; Sleep quality; Health-related Quality of Life
MeSH Terms: conditions — Kidney Failure, Chronic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A total of 124 non-diabetic peritoneal dialysis patients will be randomly assigned to two groups in a 1:1 ratio. Patients in group A will receive NCPD from Week 1 to Week 12 and then switch to CAPD from Week 13 to Week 24. Patients in group B will receive CAPD treatment from Week 1 to Week 12 and then switch to NCPD from Week 13 to Week 24.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nocturnal Continuous Cyclical Peritoneal Dialysis (NCPD) (Experimental): In NCPD, patients uses a machine to exchange fluid to perform dialysis at night.
  Interventions: Procedure: Group A and Group B
- Continuous Ambulatory Peritoneal Dialysis (CAPD) (Active Comparator): In CAPD, patients perform dialysis with manual fluid change at daytime .
  Interventions: Procedure: Group A and Group B

INTERVENTIONS:
Procedure: Group A and Group B — Group A: Participants receive NCPD for 12 weeks and then switch to CAPD for another 12 weeks.Group B: Participants receive CAPD for 12 weeks and then switch to NCPD for another 12 weeks.
  Arms: Nocturnal Continuous Cyclical Peritoneal Dialysis (NCPD)
Procedure: Group A and Group B — Group A: Participants receive NCPD for 12 weeks and then switch to CAPD for another 12 weeks.Group B: Participants receive CAPD for 12 weeks and then switch to NCPD for another 12 weeks.
  Arms: Continuous Ambulatory Peritoneal Dialysis (CAPD)

SUMMARY:
Background: Compared with continuous ambulatory peritoneal dialysis (CAPD), nocturnal continuous cyclic peritoneal dialysis (NCPD) uses a machine to exchange fluid to perform dialysis at night, allowing patients to work or study normally during daytime. Since the dialysis fluid retention time of NCPD patients is shorter than that of CAPD, this RCT was designed to investigate whether there is a difference in the efficacy between the two modalities on peritoneal dialysis.

Design: Randomized, open-label, cross-over, multi-center clinical trial.

Objective:

Primary Objective: To compare the adequacy of peritoneal dialysis between NCPD and CAPD in non-diabetic patients.

Secondary Objective: To compare the effects of NCPD and CAPD on the quality of life, including sleep quality, nocturnal blood pressure, and ultra-filtration volume in non-diabetic patients.

Hypothesis: In non-diabetic patients, NCDP is non-inferior to CAPD in peritoneal dialysis adequacy.

Methods: A total of 124 non-diabetic peritoneal dialysis patients will be enrolled and randomly assgined into two groups in a 1:1 ratio. Patients in group A will receive NCPD treatment from 1 to 12 weeks and then switch to CAPD treatment from 13 to 24 weeks, while patients in group B will receive CAPD treatment from 1 to 12 weeks and then switch to NCPD treatment from 13 to 24 weeks. All patients are required to sign an informed consent before enrollment. The enrolled patients are planned to be followed every 4 weeks, and unplanned visits will be arranged if necessary. The peritoneal dialysis adequacy (weekly total Kt/V) of the patients will be assessed at baseline and at the corresponding visit points. The average daily ultra-filtration volume during the two modalities of treatment will be compared. Sleep quality parameters will be collected using a contact-free continuous vital signs monitoring equipment at baseline, Week 12 and Week 24. The health-related quality of life and social function will be analyzed using the Kidney Disease Quality of Life 36-item short form survey (KDQOL-36) and Social Disability Screening Schedule (SDSS) questionnaire. Twenty-four-hour Ambulatory Blood Pressure (ABP) will be monitored at baseline, Week 12, and Week 24.

DETAILED DESCRIPTION:
Sample Size Estimation:

Clinical data from previous studies showed that the total weekly Kt/V of non-diabetic peritoneal dialysis patients was 2.4 (95% CI: 1.46-3.38), the change in Kt/V after 3 months of treatment was -0.02 (95% CI: -0.64-0.59), and the standard deviation of the change was 0.31 (95% CI: 0.26-0.36). Based on the above data, we estimated the sample size.

For the primary efficacy outcome (the difference of Kt/V score between NCPD and CAPD patients), the non-inferiority test shows that 110 patients could provide 90% power to detect an absolute difference of 0 when the margin of non-inferiority is 0.1 with a common standard deviation of 0.36 at one-sided significance level α=0.025. Considering the 10% rate of loss to follow-up, 124 cases (62 cases in each sequence) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years;
2. Maintenance peritoneal dialysis for ≥ 1 month;
3. Weekly total CrCL ≥ 45 liters/week/1.73m2 body surface area;
4. Total weekly Kt/V ≥ 1.7.

Exclusion Criteria:

1. Patients with diabetes mellitus;
2. Maintained peritoneal dialysis solution with a glucose concentration >2.5%;
3. Combined with acute events of cardiovascular disease(CVD), cardiac function ≥ New York Heart Association (NYHA) class III;
4. Episodes of peritonitis in the past 1 month;
5. Abdominal surgery other than PD catheter insertion in the past 3 months;
6. Planned kidney transplant in the last 6 months;
7. Active hepatitis, cirrhosis, psychiatric disease, malignancy, pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Total Weekly Kt/V | Week 0, 4, 8, 12, 16, 20, and 24
  Total weekly Kt/V will be detected at baseline and every visit point (Week 0, 4, 8, 12, 16, 20, and 24). The mean total weekly Kt/V score during NCPD treatment will be compared with that of CAPD.
  Standardized formula will be used to calculate total weekly Kt/V score: Kt/V = Kd×T/V. Kd is peritoneal urea nitrogen removal rate. T is the time (unit: min). V represents the urea distribution volume (weight×0.58).

SECONDARY OUTCOMES:
Sleep Quality | Week 12, and 24
  Sleep quality will be monitored by a contact-free continuous vital signs monitoring equipment at Week 12 and Week 24. Total sleep duration, time required to fall asleep, duration and proportion of deep/light sleep/REM phases, awake duration, and number of body movements will be reported after sleep monitoring.
Health-related Quality of Life and Social Function | Week 0, 12, and 24
  Kidney Disease Quality of Life Short Form 36 (KDQOL-36), a self-reported questionnaire, will be assessed at baseline, Week 12, and Week 24. The total scores will be calculated to evaluate the health-related quality of life at every module after transformed raw scores linearly to a range of 0 (minimum value) to 100 (maximum value) .
  Social Disability Screening Schedule (SDSS) questionnaire will be assessed at baseline, Week 12, and Week 24. The total score will be calculated to evaluate the social function.
Ambulatory Blood Pressure (ABP) | Week 0, 12, and 24
  Twenty-four-hour ABP will be monitored at baseline, Week 12, and Week 24, including daytime average blood pressure, nocturnal average blood pressure, and blood pressure variability.
Peritoneal Ultrafiltration Volume (UV) | Everyday during treatment
  Peritoneal UV will be recorded daily during treatment. The average peritoneal UV will be compared between the two modalities.
  Net ultrafiltration volume will be calculated as the volume of the drained dialysate (L) minus the volume of infused dialysis fluid (L).

CONTACTS AND LOCATIONS:
Overall Officials: Fanfan Hou, MD,PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
During the study period, individual participant data (IPD) is shared between the sponsor and collaborators. After the study is completed, IPD is available to other researchers on the condition of obtaining consent from the principal investigator.

REFERENCES:
- [Background] Guo A, Mujais S. Patient and technique survival on peritoneal dialysis in the United States: evaluation in large incident cohorts. Kidney Int Suppl. 2003 Dec;(88):S3-12. doi: 10.1046/j.1523-1755.2003.08801.x. PMID 14870873
- [Background] Li PK, Chow KM, Van de Luijtgaarden MW, Johnson DW, Jager KJ, Mehrotra R, Naicker S, Pecoits-Filho R, Yu XQ, Lameire N. Changes in the worldwide epidemiology of peritoneal dialysis. Nat Rev Nephrol. 2017 Feb;13(2):90-103. doi: 10.1038/nrneph.2016.181. Epub 2016 Dec 28. PMID 28029154
- [Background] Bieber SD, Burkart J, Golper TA, Teitelbaum I, Mehrotra R. Comparative outcomes between continuous ambulatory and automated peritoneal dialysis: a narrative review. Am J Kidney Dis. 2014 Jun;63(6):1027-37. doi: 10.1053/j.ajkd.2013.11.025. Epub 2014 Jan 11. PMID 24423779
- [Background] Rabindranath KS, Adams J, Ali TZ, Daly C, Vale L, Macleod AM. Automated vs continuous ambulatory peritoneal dialysis: a systematic review of randomized controlled trials. Nephrol Dial Transplant. 2007 Oct;22(10):2991-8. doi: 10.1093/ndt/gfm515. Epub 2007 Sep 17. PMID 17875571
- [Background] Roumeliotis A, Roumeliotis S, Leivaditis K, Salmas M, Eleftheriadis T, Liakopoulos V. APD or CAPD: one glove does not fit all. Int Urol Nephrol. 2021 Jun;53(6):1149-1160. doi: 10.1007/s11255-020-02678-6. Epub 2020 Oct 13. PMID 33051854
- [Background] Beduschi Gde C, Figueiredo AE, Olandoski M, Pecoits-Filho R, Barretti P, de Moraes TP; all centers that contributed to the BRAZPD. Automated Peritoneal Dialysis Is Associated with Better Survival Rates Compared to Continuous Ambulatory Peritoneal Dialysis: A Propensity Score Matching Analysis. PLoS One. 2015 Jul 27;10(7):e0134047. doi: 10.1371/journal.pone.0134047. eCollection 2015. PMID 26214801
- [Background] Jung HY, Jang HM, Kim YW, Cho S, Kim HY, Kim SH, Bang K, Kim HW, Lee SY, Jo SK, Lee J, Choi JY, Cho JH, Park SH, Kim CD, Kim YL; EQLIPS Study Group. Depressive Symptoms, Patient Satisfaction, and Quality of Life Over Time in Automated and Continuous Ambulatory Peritoneal Dialysis Patients: A Prospective Multicenter Propensity-Matched Study. Medicine (Baltimore). 2016 May;95(21):e3795. doi: 10.1097/MD.0000000000003795. PMID 27227956
- [Background] Michels WM, van Dijk S, Verduijn M, le Cessie S, Boeschoten EW, Dekker FW, Krediet RT; NECOSAD Study Group. Quality of life in automated and continuous ambulatory peritoneal dialysis. Perit Dial Int. 2011 Mar-Apr;31(2):138-47. doi: 10.3747/pdi.2010.00063. Epub 2011 Feb 28. PMID 21357936
- [Background] Cortes-Sanabria L, Paredes-Cesena CA, Herrera-Llamas RM, Cruz-Bueno Y, Soto-Molina H, Pazarin L, Cortes M, Martinez-Ramirez HR. Comparison of cost-utility between automated peritoneal dialysis and continuous ambulatory peritoneal dialysis. Arch Med Res. 2013 Nov;44(8):655-61. doi: 10.1016/j.arcmed.2013.10.017. Epub 2013 Nov 8. PMID 24211750
- [Derived] Driehuis E, Eshuis M, Abrahams A, Francois K, Vernooij RW. Automated peritoneal dialysis versus continuous ambulatory peritoneal dialysis for people with kidney failure. Cochrane Database Syst Rev. 2024 Sep 11;9(9):CD006515. doi: 10.1002/14651858.CD006515.pub2. PMID 39258519